CLINICAL TRIAL: NCT06140602
Title: Postprandial Urolithin Response to a Pecan-Enriched Meal
Brief Title: Postprandial Urolithin Patterns Following Pecan Consumption
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Georgia (Other)
Collaborators: Georgia Commodity Commission for Pecans (Unknown); American Pecan Counsel (Unknown)
Responsible Party: Principal Investigator, Chad Paton, Associate Professor, Principal Investigator Chad M. Paton, PhD, University of Georgia
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Health Services Research
Other Study IDs: PROJECT00007260
Record Dates: First submitted 2023-11-14; First posted 2023-11-20 (Actual); Last update posted 2023-11-24 (Actual); Status verified 2023-11

CONDITIONS: Change in Plasma Urolithins and Vitamin E
Keywords: Urolithins; Pecans; Dietary biomarker; Tocopherols

STUDY DESIGN:
Intervention Model Description: Randomized, crossover, single-blinded study with one intervention (breakfast milkshake
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention shake (Experimental): The pecan shake is comprised of 1% milk, chocolate powder (Nesquik), soy lecithin, whole blended pecans, and water.
  Interventions: Other: Intervention shake
- Control shake (No Intervention): the control cream shake is comprised of 1% milk, chocolate powder (Nesquik), soy lecithin, dextrin, heavy whipping cream, and water.

INTERVENTIONS:
Other: Intervention shake — The pecan shake contains 69g of pecans
  Other Names: Pecan shake
  Arms: Intervention shake

SUMMARY:
Pecan-enriched diets have been linked to improved cardiovascular health, including postprandial blood lipids and microvascular reactivity in older adults. This has led to recommendations to increase regular pecan consumption, however there is no consistent plasma measure of pecan intake. Traditionally, plasma tocopherols have been used, although they reach peak concentrations in plasma around 6-8 hours post pecan consumption, leading to high variability at 24 hours. Therefore, a more reliable biomarker of pecan consumption needs to be defined. The purpose of this study is to analyze the postprandial response of urolithins in human plasma after a pecan enriched meal and compare their appearance pattern to tocopherols. This single blind, randomized crossover trial is designed to provide two acute meal challenges for each participant (anticipated n=30, BMI 18.5 - 24.9, age 18-30y) with a washout period of ~14 days between each challenge. The intervention meal contains 68g of pecans and the control shake contains whipped cream instead of pecans, and the order of each meal will be randomly assigned. Blood draws will be collected at fasting (0-h) and every 2 hours until 8 hours postprandial, then at 12-, 24-, and 48h after the meal. The levels of urolithins and tocopherols will be quantified through liquid chromatography tandem mass spectrometry. To our knowledge, this is the first time urolithins will be tracked in plasma up to 48h post meal. This study will be used to establish of a new and more consistent dietary biomarker for pecans.

DETAILED DESCRIPTION:
This study aims to find a new marker for the consumptions of pecans, and any other food containing ellagitannins. Our goal is to find out the patterns of Urolithins (Uros), a metabolite originated from ellagic acid by the gut microbiota. Previous study supports that Urolithins and it's glucuronides conjugates, especially Uro A glucuronide, increase in blood plasma after 4-week intervention of chronic consumption of pecans. However, little is known about Uros in plasma after an acute meal containing ellagitannins. For this reason, this project's goal is to be able to hourly track Uros after a pecan enriched meal.This trial will be a double-blinded, randomized, cross-over design in humans. There will be three study visits. The screening visit (v1) will entail signing informed consent documents, anthropometric measurements, and receiving their dinner entrée for the night before v2. The two testing visits (v2 and v3) include blood draws after consuming one of the two different test meals: 1) a breakfast shake consisting primarily of pecans, Nesquik and 1% milk, or 2) a breakfast shake consisting primarily of heavy whipping cream, Nesquik and 1% milk. There will be a 6-14 day washout period between each study visit. There will be a total of thirty participants in this study (n=30). All visits will take place in the Human Nutrition Lab (HNL) at the University of Georgia in Athens.

Only Dr. Chad Paton and/or members of his research team will screen potential participants interested in the study. The screening process will be done over the phone, or in person. In contrast, the consent process will be done in person only. If potential participants complete an online interest screening form they will be contacted by the researchers listed above. These researchers will conduct the full telephone screening and inform the potential participant whether or not they qualify for the study. For participants that have completed the online interest form, researchers will clarify questions that have previously been asked, and focus on collecting new information in order to compete the full screening. If the potential participant does qualify for the study, an in-person Screening and Consent Visit (v1) will be scheduled during or after this phone call.

During the in-person Screening and Consent Visit, the participant will be provided with detailed verbal and written information regarding the study and activities it entails. This includes information regarding the nutritional content of the breakfast shakes, pre-visit 24-hour diet protocol (verbal and paper-copy instructions), and blood drawing procedures. If the participant willingly consents to the study and signs the consent form, the investigators will proceed with the rest of the screening visit. If participants are eligible to participate in the study after the Screening Visit, then they will complete two additional testing visits. After the fasting blood draw, participants will be given a breakfast shake to consume. Liquid chromatography tandem mass spectrometry (LC-MS/MS) will be used to quantify plasma urolithin-A, -B, and -C as well as their glucuronide conjugates. Additionally, LC-MS/MS will be used to measure plasma tocopherols and tocotrienols. Plasma changes in triglycerides and glucose will be determined by enzyme assay.

ELIGIBILITY:
Inclusion Criteria:

* Healthy individuals with BMI between 18.5 - 29.9 kg/m2
* Does not make use of medication (Birth control, and antidepressants SSRIs accepted)
* Does not make use of any nicotine products
* Has not been diagnosed with any diseases that can impair swallowing, digestion or lipid metabolism

Exclusion Criteria:

* Individuals with BMI < 18.5 or BMI > 29.9 kg/m2
* Individuals with chronic diseases of the gastrointestinal system
* Individuals currently taking antibiotics or any other medications not included on the inclusion criteria
* Individuals that have a current fever, or have any infection
* Individuals can not be taking prebiotics/probiotics supplementation, as well as multivitamin.

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-07-18 (Actual); Primary Completion 2024-05-30 (Estimated); Study Completion 2024-07-30 (Estimated)

PRIMARY OUTCOMES:
Urolithins pattern in blood plasma | baseline blood draw 8 hours postprandial, then at 12 hours, 24 hours and 48 hours postprandial time points
  A fasting/baseline blood draw, followed to 2 hours, 4 hours, 6 hours, 8 hours, 12 hours 24h, 48h.

SECONDARY OUTCOMES:
Which isoform of Uros (A, B, C and it's glucuronides (Uro A-G, Uro B-G) will peak | baseline blood draw 8 hours postprandial, then at 12 hours, 24 hours and 48 hours postprandial time points
  Which isoform will be seeing in greater amount when tracked

CONTACTS AND LOCATIONS:
Overall Officials: Chad M Paton, PhD, Principal Investigator — University of Georgia
Locations (1):
- Human Nutrition Lab, Athens, Georgia, United States

IPD SHARING:
Plan to Share IPD: No